CLINICAL TRIAL: NCT03766334
Title: Efficacy and Safety of Highland Barley Diet on Glucose Variability in Patients With Type 1 Diabetes Mellitus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project closure
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xuefeng Yu, Chief of Department of Endocrinology, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-T1DM-CGM-001
Record Dates: First submitted 2018-07-02; First posted 2018-12-06 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Highland Barley Diet; Glucose variability

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Diet+Highland Barley Diet (Experimental): Diabetes Diet+Highland Barley Diet(20g, thrice-daily)
  Interventions: Dietary Supplement: Highland Barley Diet
- Diabetes Diet (No Intervention): only Diabetes Diet

INTERVENTIONS:
Dietary Supplement: Highland Barley Diet — Highland Barley Diet(20g, thrice-daily)
  Arms: Diabetes Diet+Highland Barley Diet

SUMMARY:
Approximately 80 patients will be enrolled in the study from China and randomized in a 1:1 ratio to one of the 2 treatment arms:diabetes diet+highland barley diet; or diabetes diet.

Study treatment will continue for 12 weeks. The primary efficacy measure is the change in MAGE from continuous glucose monitoring system at 12 weeks. The study consists of 3 periods: a 1-week screening (period A), a 8-day run-in period (period B) and a 12-week treatment period (period C). Continuous glucose monitoring system will be used in baseline and endpoint.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label comparison of the effects and safety of barley meal plus diabetes diet on blood glucose fluctuations in patients with type 1 diabetes (T1DM) using multiple daily insulin injections (MDI). , parallel test. About 80 patients with T1DM were enrolled in the preliminary trial. During the lead-in period, no interventions were given to the patient's diet from day 1 to day 4, and diabetes diet education and guidance were given from day 5 to day 8, depending on the patient's blood glucose and diet. Personalization of habits, weights, and activities, etc., establish a diabetes diet. At the end of the lead-in period, patients were randomly divided into two treatment groups according to the ratio of 1:1: Observation group: Diabetes diet + barley diet. (The barley meal group diet was formulated according to the diabetes diet, but each meal was replaced with 20g barley nutrition powder and other calories instead of part of the diet. In the control group: Diabetes diet; dietary treatment after randomization will continue for 12 weeks. From the induction period to the treatment period 6 days, treatment period 10-12 weeks

ELIGIBILITY:
Inclusion Criteria:

1. type 1 diabetes patients with disease duration more than one year
2. HbA1c ≥7.0 % and < 11.0 %
3. Men and women (non-pregnant and using a medically approved birthcontrol method) aged ≥ 18 and ≤ 65 years
4. BMI ≥ 18 and ≤ 26 kg/m2

Exclusion Criteria:

1. Type 2 diabetes or other specific types of diabetes
2. Pregnancy, preparation for pregnancy, lactation and women of childbearing age incapable of effective contraception methods
3. Uncooperative subject because of various reasons
4. Abnormal liver function, glutamic-pyruvic transaminase (ALT) and glutamic-oxaloacetic transaminase (AST) > twice the upper limits of normal
5. Impairment of renal function, serum creatinine: ≥ 133mmol/L for female，≥ 135mmol/L for male
6. Serious chronic gastrointestinal diseases
7. Edema
8. Serious heart diseases, such as cardiac insufficiency (level III or more according to NYHA), acute coronary syndrome and old myocardial infraction
9. Blood pressure: Systolic blood pressure (SBP) ≥ 180mmHg and/or diastolic blood pressure (DBP) ≥ 110mmHg
10. White blood count (WBC) < 4.0×109/L or platelet count (PLT) < 90×109/L，or definite anemia (Hb：< 120g/L for male, < 110g/L for female), or other hematological diseases
11. Endocrine system diseases, such as hyperthyroidism and hypercortisolism
12. Experimental drug allergy or frequent hypoglycemia
13. Psychiatric disorders, drug or other substance abuse
14. Diabetic ketoacidosis and hyperosmolar nonketotic coma requiring insulin therapy
15. Stressful situations such as surgery, serious trauma and so on
16. Chronic hypoxic diseases such as pulmonary emphysema and pulmonary heart disease
17. Combined use of drugs effecting glucose metabolism such as glucocorticoid Tumor, especially bladder tumor and/or family history of bladder tumor and/or long-term hematuria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Average blood glucose fluctuations at endpoint and baseline | from baseline to 12-week endpoint
  Objective to investigate the effect of combination diabetes diet and highland barley diet on glucose variability in insufficient control patients with type 1 diabetes.

SECONDARY OUTCOMES:
Glycated hemoglobin(endpoint)-Glycated hemoglobin(baseline) | from baseline to 12-week endpoint
  Objective to investigate the effect of combination diabetes diet and highland barley diet on glucose control in patients with type 1 diabetes.
insulin dose(endpoint)-insulin dose(baseline) | from baseline to 12-week endpoint
  Objective to investigate the effect of combination diabetes diet and highland barley diet on insulin dose in patients with type 1 diabetes.
Quality of life assessment scale SF-36(endpoint)-Quality of life assessment scale SF-36(baseline) | from baseline to 12-week endpoint
  Objective to investigate the effect of combination diabetes diet and highland barley diet on life quality in patients with type 1 diabetes.
Body mass index(endpoint)-Body mass index(baseline) | from baseline to 12-week endpoint
  Objective to investigate the effect of combination diabetes diet and highland barley diet on BMI in patients with type 1 diabetes.
beta-cell function at endpoint and baseline | from baseline to 12-week endpoint
  Objective to investigate the effect of combination diabetes diet and highland barley diet on beta-cell function in patients with type 1 diabetes.
Waist circumference(endpoint)-Waist circumference(baseline) | from baseline to 12-week endpoint
  Objective to investigate the effect of combination diabetes diet and highland barley diet on waist circumference in patients with type 1 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: xuefeng Yu, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No